CLINICAL TRIAL: NCT03233516
Title: Trial of Respiratory Infections in Children for Enhanced Diagnostics
Acronym: TREND
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm South General Hospital (Other); Science for Life Laboratory (Unknown); Uppsala University (Other); Astrid Lindgren Children´s Hospital (Other); Sahlgrenska University Hospital (Other); Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Tobias Alfvén, Associate professor, Karolinska Institutet
Other Study IDs: 2017/958-31
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Community-acquired Pneumonia
Keywords: Community-acquired pneumonia; Pediatrics; Etiology; Point-of-care test; MxA; CRP; Procalcitonin; Infectious diseases; Respiratory viruses; Pediatric asthma
MeSH Terms: conditions — Community-Acquired Pneumonia; Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — * capillary lithium-heparin tube (will be separated into two aliquots and diluted in a commercial buffer)
  * capillary point-of-care test CRP
  * nasopharyngeal swab for Mari-POC (diluted in 1.3ml MariPOC RTI buffer)
  * nasopharyngeal aspirate (diluted into 1.3ml saline) divided into three aliquots:
    1. Real-time PCR-analysis of respiratory agents (400μl)
    2. Frozen down at -80°C for study IV (400μl)
    3. Available for routine microbiological testing as ordered by the attending physician. If not used, frozen down at -80°C for potential reanalyses. (500μl)
  All samples will be taken within 24h from arrival at the emergency unit and time for both blood and nasopharynx samples will be registered. It will also be noted if antibiotics have been given before samples taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases with clinical CAP: Children 1-59 months at Sachs' Children and Youth Hospital with clinical CAP (both severe and non-severe) according to WHO-criteria.
- Control subjects: Children 1-59 months at Sachs' Children and Youth Hospital treated for a minor orthopedic (elective (e.g. hand surgery) or acute) or minor surgical disease, e.g. minor trauma (excluding e.g. appendicitis, major burns, major trauma).

SUMMARY:
The overall aim of the TREND study is to improve the differential diagnosis of bacterial and viral etiology in children below 5 years of age with clinical community acquired pneumonia.

Specific objectives:

* To assess the diagnostic accuracy of MxA for viral CAP (sub-study I)
* To study etiologies in children with CAP (sub-study II)
* To evaluate sensitivity and specificity for MariPOC® Respi test versus PCR for detection of respiratory viruses (sub-study III)
* To assess sensitivity and specificity for a novel RPA-based point-of-care test versus PCR for detection of respiratory viruses (sub-study IV)
* To assess long-term complications in children with CAP (sub-study V

The study takes place at Sachs' Children and Youth hospital in Stockholm.

DETAILED DESCRIPTION:
Background: Respiratory viral and bacterial infections are hard to distinguish clinically, and many children with viral infections receive unnecessary treatment with antibiotics, which contributes to development and spread of antibiotic resistance. Therefore, there is a need for new point-of-care diagnostic tests that better distinguish viral from antibiotic-requiring bacterial infections, particularly in children presenting with suspected clinical community-acquired pneumonia (CAP), and thus assist health-care workers decision making and improve rational use of antibiotics.

Myxovirus resistance protein A (MxA) is a promising biomarker for viral infection, but no studies have investigated MxA in children with CAP. Procalcitonin (PCT) is used as a biomarker for severe bacterial infection as the protein rapidly increases in plasma levels in response to stress and systemic infection. PCT has been reported to be more specific for bacterial infection as compared to CRP, but there are conflicting data on the clinical utility of PCT in children with CAP.

The role of viruses and atypical bacteria in childhood CAP Is increasingly recognized. Recent studies have reported an increasing incidence of B. pertussis and there have been several deaths in previously healthy infants associated with whooping cough in Sweden over the last ten years. Consequently, there is a need for new etiologic studies in childhood CAP.

Real-time PCR is currently considered gold-standard for detection of respiratory viruses in children with respiratory tract infection. Nevertheless, the turn-around time is usually long and the test results can rarely be used for decision making regarding treatment. There are currently several new antigen-based point-of-care tests of respiratory infections on the market, one is Multianalyte Point-of-care Antigen Detection Test System (MariPOC®) Respi. The sensitivity for respiratory syncytial virus (RSV) and influenza virus is as high as 90% as compared to PCR, the current gold-standard PCR, but, the sensitivity for less common respiratory viruses such as metapneumovirus (hMPV), parainfluenza virus (PIV), coronavirus and bocavirus have been insufficiently investigated.

Recombinase polymerase amplification (RPA) is a nucleic acid amplification method that doesn't require thermal cycling. As the test reaction can be carried out at room temperature it is a particularly interesting method for resource-limited settings where the need for new diagnostic tests is high.

Studies on long-term outcomes of radiologically confirmed bacterial CAP have indicated that the disease is associated with later development of asthma and decreased lung-function. Given the ongoing change in etiology of pediatric CAP, there is a need for new studies of long-term complications in pediatric CAP.

Overall Aim:

The overall aim of the TREND study is to improve the differential diagnosis of bacterial and viral etiology in children below 5 years of age with clinical CAP.

Specific objectives:

* To assess the diagnostic accuracy of MxA for viral CAP (sub-study I)
* To study etiologies in children with CAP (sub-study II)
* To evaluate sensitivity and specificity for MariPOC® Respi test versus PCR for detection of respiratory viruses (sub-study III)
* To assess sensitivity and specificity for a novel RPA-based point-of-care test versus PCR for detection of respiratory viruses (sub-study IV)
* To assess long-term complications in children with CAP (sub-study V)

Study Design:

The TREND study is a hospital-based prospective observational study of children with clinical CAP with asymptomatic controls at the emergency department at Sachs' Children and Youth hospital, Stockholm.

Case definition Children 1-59 months with clinical CAP according to WHO-criteria.

Bronchodilator challenge:

Inhalation with a rapid acting bronchodilator will be administered to children with wheezing and in-drawings to improve the specificity of the WHO clinical CAP criteria as suggested by the PERCH study team. Resolved in-drawings after bronchodilator challenge will be recorded but not considered an exclusion criteria to be able to exclude these patients in a sub-analysis.

Control definition:

Children 1-59 months at Sachs' Children and Youth Hospital treated for a minor orthopedic or minor surgical disease. The parents to the controls will be contacted via email/telephone 1-2 weeks after enrollment and be asked whether the child has developed respiratory symptoms or not. No matching will be performed but adjustments for age and season will be performed in the analyses.

Sampling:

A capillary blood sample and nasopharyngeal swabs/aspirates will be collected from all study subjects.

Microbiological and Biochemistry Analyses:

MariPOC® Respi as well as real-time PCR analysis (detecting: 16 respiratory viruses as well as Streptococcus pneumoniae, Bordetella pertussis, B. parapertussis and Mycoplasma pneumoniae) will be performed.

Biochemistry Analyses:

Serum MxA, procalcitonin and CRP levels will be analysed.

Study Variables:

Information regarding the study subject, number of siblings, days of illness, current symptoms, vaccinations, antibiotic treatment, medication, underlying diseases, heredity for asthma, previous hospitalization, recent stay abroad, allergies, smoking, recent travel abroad, recent contact with unwell individual, breastfeeding, preschool, origin of parents and socio-economic status will be collected through a standardized questionnaire based on previous studies.

Clinical parameters will be registered by the study doctor responsible for patient screening/enrolment in line with the study protocol of PERCH. Some of the clinical parameters included in the PERCH protocol are very rare in a Swedish context and to avoid overloading of the case report form, these will not be systematically registered at inclusion. However, information about these symptoms will be retrospectively collected from the medical records. Some clinical parameters are routinely recorded multiple times at the emergency unit. In these cases, the most extreme value (highest pulse/respiratory rate/body temperature/etc and lowest peripheral oxygen saturation) during the visit at the emergency unit until enrolment will be recorded. Information regarding admission, length of stay, radiological, routine clinical examination, microbiological and chemistry analyses, treatment, discharge diagnosis and complications will be retrospectively collected from the medical records.

All study subjects will be linked to the National Vaccination register to collect information regarding previous immunizations. To allow assessment of long-term complication, study subjects will also be linked to the National Patient Register, the National Death Register and the National Prescribed Drug Register for collection of discharge diagnoses according to ICD-10 as well as prescribed drugs.

Classification of Disease:

Etiology will be classified as probable or definitive based on clinical significance of the different microbiological test in the studies above. In TREND, the combination of probable and definitive etiology will be used in the main analysis, whereas children with definitive etiology will be assessed separately in a sub-analysis.

Definitive Viral Infection:

• PCR positive for influenza, RS virus, metapneumovirus or parainfluenza virus

Probable Viral Infection:

* PCR positive for adenovirus
* PCR positive for coronavirus, rhinovirus, bocavirus or enterovirus AND CRP <20 AND reported fever >24h.

Definitive Bacterial Infection:

* positive bacterial blood culture in blood or pleura fluid
* positive pneumococcal antigen test in pleura fluid

Probable Bacterial Infection:

* CRP >80 (children ≤2 years) / >120 (children 2-5 years) AND/OR
* Radiographic evidence of empyema on X-ray or ultrasound AND/OR
* Large dense infiltrate or lobar consolidation on chest x-ray

Definitive Atypical Bacterial Infection:

• Positive PCR B. pertussis or B. parapertussis

Probable Atypical Bacterial Infection:

• Positive PCR M. pneumoniae

Undetermined:

• Cases not fulfilling any criteria above

Mixed Viral-bacterial Infection:

• Children fulfilling criteria for both viral and bacterial infection

Classification of Long-term Complications:

Long-term complications (asthma and number of hospital-requiring respiratory infections) will be assessed after 3, 7 and 10 years following study completion by linking to the National Patient Register. Asthma will be classified as ICD-10 diagnosis of J45 or ≥3 prescriptions of inhalation steroids, beta-2-agonists or leukotriene antagonists according to the Prescribed Drug Register.

Power Calculation:

For the sample size calculation, the investigators focused on the assessment of MxA-levels in cases with viral CAP as compared to cases with bacterial CAP/controls (study I). Two power calculations were made, one for viral CAP versus bacterial CAP and one for viral CAP versus controls. The following assumptions were made:

A difference in MxA-level of 500µg/l between the groups was considered clinically relevant. A standard deviation of 1000 and 300 was assumed in cases with viral CAP and bacterial CAP/controls respectively based on previous studies on MxA.

Using an alpha-level of 0.05 (two-sided) at an 80% power, with an additional 20% addition to account for non-parametric testing and multivariate analyses, 42 children in each group (viral CAP, bacterial CAP and controls) would be needed.

To ensure that enough of the included cases would fulfill the TREND definition of viral and bacterial CAP, the proportion of viral respectively bacterial CAP (TREND definition) was calculated in our previous study that assessed Swedish children with x-ray verified CAP. By doing this, the prevalence of viral and bacterial CAP was estimated to 45% and 14% respectively. Hence 300 cases and 42 controls would be needed to ensure sufficient collection of cases with viral and bacterial CAP respectively. The investigators also would like to compare cases with viral CAP with controls testing positive for one or more virus by PCR. In our previous study, 35.4% of asymptomatic children tested positive for one or more virus. To include a sufficient number of virus-positive controls, the investigators hence aim at including 300 cases and 119 controls (42/0.354=119) in the TREND-study.

Ethical Considerations:

The study will be conducted in accordance with the latest version of The Declaration of Helsinki and the fundamental principles of respect for the individual (Article 8), their right to self-determination and the right to make informed decisions (Articles 20, 21 and 22) regarding participation in research, both initially and during the course of the research.

Significance:

The findings from the TREND project can be an important step to improve the care of children with clinical CAP. Improved near-patient differential diagnosis is a prerequisite for rational antibiotic use and decreasing unnecessary antibiotic treatment. Further better diagnosis of the pathogens causing acute respiratory infections makes it easier to give advice to parents on how their children should be cared for and better surveillance in the society.

ELIGIBILITY:
Inclusion Criteria:

Cases:

(all inclusion criteria to be met to be eligible for participation in the study).

* Age 28 days to 59 months
* Reported and/or observed breathing troubles OR cough
* Observed age-adjusted tachypnea (≥50 breaths/min in children 1-12 months, ≥40/min in children >1year) OR chest in-drawings
* Written informed consent

Controls:

(all inclusion criteria to be met to be eligible for participation in the study).

* Age 28 days to 59 months
* Minor surgical or orthopedic disease (elective (e.g. hand surgery) or acute) or minor surgical disease, e.g. minor trauma (excluding e.g. appendicitis, major burns, major trauma)
* Written informed consent

Exclusion Criteria:

Cases:

* Previously included as case in the study
* Hospitalized during last 14 days

Controls:

Symptoms of respiratory disease 7 days before enrollment

* Previously included as control in the study
* Hospitalized during last 14 days

Ages: 28 Days to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Case definition:
  Children 1-59 months at Sachs' Children and Youth Hospital with clinical CAP (both severe and non-severe) according to WHO-criteria
  Control definition:
  Children 1-59 months at Sachs' Children and Youth Hospital treated for a minor orthopedic (elective (e.g. hand surgery) or acute) or minor surgical disease, e.g. minor trauma (excluding e.g. appendicitis, major burns, major trauma). No matching will be performed but adjustments for age and season will be performed in the analyses.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
MxA - cases with viral and bacterial clinical CAP | 2021
  Clinically relevant difference in MxA-levels between cases with viral and bacterial clinical CAP
Mxa viral clinical CAP and controls | 2021
  Clinically relevant difference in MxA-levels between cases with viral clinical CAP and controls
PCR - respiratory pathogens in cases and controls | 2020
  Proportion of respiratory pathogens in cases and controls, using real time PCR
Sensitivity and specificity - MariPOC | 2021
  Sensitivity and specificity for different respiratory viruses with MariPOC® Respi as compared to real-time PCR
Sensitivity and specificity a novel PCR-based point-of-care test | 2021
  Sensitivity and specificity for different respiratory viruses with a novel PCR-based point-of-care test as compared to PCR
Difference asthma prevalence and number of hospital-requiring respiratory infections - cases and controls, | 2027
  Difference in asthma prevalence between cases and controls and difference in number of hospital-requiring respiratory infections between cases and controls after 3, 7 and 10 years

SECONDARY OUTCOMES:
Specific assessment of MxA as a clinical biomarker | 2021
  Clinically relevant difference in MxA-levels comparing cases with viral clinical CAP with cases with atypical and mixed viral-bacterial clinical CAP as well as with controls with and without presence of respiratory viruses by PCR
Specific assessment of MxA as a clinical biomarker | 2021
  Clinically relevant differences in MxA-levels in cases with regard to specific respiratory agents
Specific assessment of MxA as a clinical biomarker | 2021
  Sensitivity and specificity for MxA in identifying viral clinical CAP
Specific assessment of MxA as a clinical biomarker | 2021
  Sensitivity and specificity for identifying viral and bacterial infection respectively for CRP, PCT and combination test of CRP, PCT and MxA
Assessment of PCT and CRP as clinical biomarkers | 2021
  Difference in CRP and PCT between children with viral, bacterial, atypical bacterial and mixed viral-bacterial infection
Descriptive statistics of study cohort with regard to etiologic agent | 2020
  Differences in symptom, antibiotic treatment, acute complications, radiologic exams admission rate and length of stay between cases with viral, bacterial, atypical bacterial and mixed viral-bacterial infection
Evaluation of MariPOC® Respi in a clinical setting | 2022
  Differences in symptom, antibiotic treatment, acute complications, radiologic exams admission rate and length of stay between cases who tested positive for respiratory virus by MariPOC® Respi as compared to those with a negative test
Assessment of long-term outcomes of children with CAP | 2027
  Number of hospital-requiring respiratory infections in cases and controls
Assessment of long-term outcomes of children with CAP | 2027
  Difference in asthma prevalence between cases with viral and bacterial clinical CAP as compared to an estimate of the prevalence in the general population
Assessment of long-term outcomes of children with CAP | 2027
  Difference in proportion of hospital-requiring respiratory infections between cases with viral, bacterial, atypical and mixed viral-bacterial infection
Evaluation of MariPOC® Respi | 2022
  Difference in MxA-levels between PCR+/MariPOC® Respi+ and PCR+/MariPOC® Respi- study subjects.
Etiology of cases in TREND study | 2020
  Estimation of etiology of cases using two levels of certainty (definitive as well as probable definition).

CONTACTS AND LOCATIONS:
Locations (1):
- Sachs' Children and Youth Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adams PF, Hendershot GE, Marano MA; Centers for Disease Control and Prevention/National Center for Health Statistics. Current estimates from the National Health Interview Survey, 1996. Vital Health Stat 10. 1999 Oct;(200):1-203. PMID 15782448
- [Background] Makela MJ, Puhakka T, Ruuskanen O, Leinonen M, Saikku P, Kimpimaki M, Blomqvist S, Hyypia T, Arstila P. Viruses and bacteria in the etiology of the common cold. J Clin Microbiol. 1998 Feb;36(2):539-42. doi: 10.1128/JCM.36.2.539-542.1998. PMID 9466772
- [Background] Elfving K, Shakely D, Andersson M, Baltzell K, Ali AS, Bachelard M, Falk KI, Ljung A, Msellem MI, Omar RS, Parola P, Xu W, Petzold M, Trollfors B, Bjorkman A, Lindh M, Martensson A. Acute Uncomplicated Febrile Illness in Children Aged 2-59 months in Zanzibar - Aetiologies, Antibiotic Treatment and Outcome. PLoS One. 2016 Jan 28;11(1):e0146054. doi: 10.1371/journal.pone.0146054. eCollection 2016. PMID 26821179
- [Background] Malhotra-Kumar S, Lammens C, Coenen S, Van Herck K, Goossens H. Effect of azithromycin and clarithromycin therapy on pharyngeal carriage of macrolide-resistant streptococci in healthy volunteers: a randomised, double-blind, placebo-controlled study. Lancet. 2007 Feb 10;369(9560):482-90. doi: 10.1016/S0140-6736(07)60235-9. PMID 17292768
- [Background] Rhedin S. Establishment of childhood pneumonia cause in the era of pneumococcal conjugate vaccines. Lancet Respir Med. 2016 Jun;4(6):423-4. doi: 10.1016/S2213-2600(16)30067-4. Epub 2016 Apr 21. No abstract available. PMID 27117546
- [Background] Reinhart K, Karzai W, Meisner M. Procalcitonin as a marker of the systemic inflammatory response to infection. Intensive Care Med. 2000 Sep;26(9):1193-200. doi: 10.1007/s001340000624. No abstract available. PMID 11089742
- [Background] Korppi M, Remes S, Heiskanen-Kosma T. Serum procalcitonin concentrations in bacterial pneumonia in children: a negative result in primary healthcare settings. Pediatr Pulmonol. 2003 Jan;35(1):56-61. doi: 10.1002/ppul.10201. PMID 12461740
- [Background] Esposito S, Tagliabue C, Picciolli I, Semino M, Sabatini C, Consolo S, Bosis S, Pinzani R, Principi N. Procalcitonin measurements for guiding antibiotic treatment in pediatric pneumonia. Respir Med. 2011 Dec;105(12):1939-45. doi: 10.1016/j.rmed.2011.09.003. Epub 2011 Sep 29. PMID 21959024
- [Background] Engelmann I, Dubos F, Lobert PE, Houssin C, Degas V, Sardet A, Decoster A, Dewilde A, Martinot A, Hober D. Diagnosis of viral infections using myxovirus resistance protein A (MxA). Pediatrics. 2015 Apr;135(4):e985-93. doi: 10.1542/peds.2014-1946. PMID 25802344
- [Background] Sambursky R, Shapiro N. Evaluation of a combined MxA and CRP point-of-care immunoassay to identify viral and/or bacterial immune response in patients with acute febrile respiratory infection. Eur Clin Respir J. 2015 Dec 10;2:28245. doi: 10.3402/ecrj.v2.28245. eCollection 2015. PMID 26672961
- [Background] Toivonen L, Schuez-Havupalo L, Rulli M, Ilonen J, Pelkonen J, Melen K, Julkunen I, Peltola V, Waris M. Blood MxA protein as a marker for respiratory virus infections in young children. J Clin Virol. 2015 Jan;62:8-13. doi: 10.1016/j.jcv.2014.11.018. Epub 2014 Nov 18. PMID 25542463
- [Background] Rhedin S, Lindstrand A, Rotzen-Ostlund M, Tolfvenstam T, Ohrmalm L, Rinder MR, Zweygberg-Wirgart B, Ortqvist A, Henriques-Normark B, Broliden K, Naucler P. Clinical utility of PCR for common viruses in acute respiratory illness. Pediatrics. 2014 Mar;133(3):e538-45. doi: 10.1542/peds.2013-3042. Epub 2014 Feb 24. PMID 24567027
- [Background] Lindstrand A, Bennet R, Galanis I, Blennow M, Ask LS, Dennison SH, Rinder MR, Eriksson M, Henriques-Normark B, Ortqvist A, Alfven T. Sinusitis and pneumonia hospitalization after introduction of pneumococcal conjugate vaccine. Pediatrics. 2014 Dec;134(6):e1528-36. doi: 10.1542/peds.2013-4177. Epub 2014 Nov 10. PMID 25384486
- [Background] Rhedin S, Lindstrand A, Hjelmgren A, Ryd-Rinder M, Ohrmalm L, Tolfvenstam T, Ortqvist A, Rotzen-Ostlund M, Zweygberg-Wirgart B, Henriques-Normark B, Broliden K, Naucler P. Respiratory viruses associated with community-acquired pneumonia in children: matched case-control study. Thorax. 2015 Sep;70(9):847-53. doi: 10.1136/thoraxjnl-2015-206933. Epub 2015 Jun 15. PMID 26077969
- [Background] Barger-Kamate B, Deloria Knoll M, Kagucia EW, Prosperi C, Baggett HC, Brooks WA, Feikin DR, Hammitt LL, Howie SR, Levine OS, Madhi SA, Scott JA, Thea DM, Amornintapichet T, Anderson TP, Awori JO, Baillie VL, Chipeta J, DeLuca AN, Driscoll AJ, Goswami D, Higdon MM, Hossain L, Karron RA, Maloney S, Moore DP, Morpeth SC, Mwananyanda L, Ofordile O, Olutunde E, Park DE, Sow SO, Tapia MD, Murdoch DR, O'Brien KL, Kotloff KL; Pneumonia Etiology Research for Child Health (PERCH) Study Group. Pertussis-Associated Pneumonia in Infants and Children From Low- and Middle-Income Countries Participating in the PERCH Study. Clin Infect Dis. 2016 Dec 1;63(suppl 4):S187-S196. doi: 10.1093/cid/ciw546. PMID 27838672
- [Background] He Q, Viljanen MK, Arvilommi H, Aittanen B, Mertsola J. Whooping cough caused by Bordetella pertussis and Bordetella parapertussis in an immunized population. JAMA. 1998 Aug 19;280(7):635-7. doi: 10.1001/jama.280.7.635. PMID 9718056
- [Background] Carlsson RM, von Segebaden K, Bergstrom J, Kling AM, Nilsson L. Surveillance of infant pertussis in Sweden 1998-2012; severity of disease in relation to the national vaccination programme. Euro Surveill. 2015 Feb 12;20(6):21032. doi: 10.2807/1560-7917.es2015.20.6.21032. PMID 25695476
- [Background] van den Brink G, Wishaupt JO, Douma JC, Hartwig NG, Versteegh FG. Bordetella pertussis: an underreported pathogen in pediatric respiratory infections, a prospective cohort study. BMC Infect Dis. 2014 Sep 30;14:526. doi: 10.1186/1471-2334-14-526. PMID 25267437
- [Background] Jartti T, Soderlund-Venermo M, Hedman K, Ruuskanen O, Makela MJ. New molecular virus detection methods and their clinical value in lower respiratory tract infections in children. Paediatr Respir Rev. 2013 Mar;14(1):38-45. doi: 10.1016/j.prrv.2012.04.002. Epub 2012 May 5. PMID 23347659
- [Background] Koskinen JO, Vainionpaa R, Meltola NJ, Soukka J, Hanninen PE, Soini AE. Rapid method for detection of influenza a and B virus antigens by use of a two-photon excitation assay technique and dry-chemistry reagents. J Clin Microbiol. 2007 Nov;45(11):3581-8. doi: 10.1128/JCM.00128-07. Epub 2007 Sep 12. PMID 17855571
- [Background] Tuuminen T, Suomala P, Koskinen JO. Evaluation of the automated multianalyte point-of-care mariPOC(R) test for the detection of influenza A virus and respiratory syncytial virus. J Med Virol. 2013 Sep;85(9):1598-601. doi: 10.1002/jmv.23660. PMID 23852685
- [Background] Sanbonmatsu-Gamez S, Perez-Ruiz M, Lara-Oya A, Pedrosa-Corral I, Riazzo-Damas C, Navarro-Mari JM. Analytical performance of the automated multianalyte point-of-care mariPOC(R) for the detection of respiratory viruses. Diagn Microbiol Infect Dis. 2015 Nov;83(3):252-6. doi: 10.1016/j.diagmicrobio.2015.07.010. Epub 2015 Jul 18. PMID 26283523
- [Background] Leblanc N, Gantelius J, Schwenk JM, Stahl K, Blomberg J, Andersson-Svahn H, Belak S. Development of a magnetic bead microarray for simultaneous and simple detection of four pestiviruses. J Virol Methods. 2009 Jan;155(1):1-9. doi: 10.1016/j.jviromet.2008.04.010. Epub 2008 Jun 2. PMID 18514335
- [Background] Chinnasamy T, Segerink LI, Nystrand M, Gantelius J, Svahn HA. A lateral flow paper microarray for rapid allergy point of care diagnostics. Analyst. 2014 May 21;139(10):2348-54. doi: 10.1039/c3an01806g. PMID 24690935
- [Background] Caliendo AM, Gilbert DN, Ginocchio CC, Hanson KE, May L, Quinn TC, Tenover FC, Alland D, Blaschke AJ, Bonomo RA, Carroll KC, Ferraro MJ, Hirschhorn LR, Joseph WP, Karchmer T, MacIntyre AT, Reller LB, Jackson AF; Infectious Diseases Society of America (IDSA). Better tests, better care: improved diagnostics for infectious diseases. Clin Infect Dis. 2013 Dec;57 Suppl 3(Suppl 3):S139-70. doi: 10.1093/cid/cit578. PMID 24200831
- [Background] Burgess JA, Abramson MJ, Gurrin LC, Byrnes GB, Matheson MC, May CL, Giles GG, Johns DP, Hopper JL, Walters EH, Dharmage SC. Childhood infections and the risk of asthma: a longitudinal study over 37 years. Chest. 2012 Sep;142(3):647-654. doi: 10.1378/chest.11-1432. PMID 22459783
- [Background] Chan JY, Stern DA, Guerra S, Wright AL, Morgan WJ, Martinez FD. Pneumonia in childhood and impaired lung function in adults: a longitudinal study. Pediatrics. 2015 Apr;135(4):607-16. doi: 10.1542/peds.2014-3060. Epub 2015 Mar 2. PMID 25733757
- [Background] Scott JA, Wonodi C, Moisi JC, Deloria-Knoll M, DeLuca AN, Karron RA, Bhat N, Murdoch DR, Crawley J, Levine OS, O'Brien KL, Feikin DR; Pneumonia Methods Working Group. The definition of pneumonia, the assessment of severity, and clinical standardization in the Pneumonia Etiology Research for Child Health study. Clin Infect Dis. 2012 Apr;54 Suppl 2(Suppl 2):S109-16. doi: 10.1093/cid/cir1065. PMID 22403224
- [Background] Brittain-Long R, Westin J, Olofsson S, Lindh M, Andersson LM. Access to a polymerase chain reaction assay method targeting 13 respiratory viruses can reduce antibiotics: a randomised, controlled trial. BMC Med. 2011 Apr 26;9:44. doi: 10.1186/1741-7015-9-44. PMID 21521505
- [Background] Almqvist C, Adami HO, Franks PW, Groop L, Ingelsson E, Kere J, Lissner L, Litton JE, Maeurer M, Michaelsson K, Palmgren J, Pershagen G, Ploner A, Sullivan PF, Tybring G, Pedersen NL. LifeGene--a large prospective population-based study of global relevance. Eur J Epidemiol. 2011 Jan;26(1):67-77. doi: 10.1007/s10654-010-9521-x. Epub 2010 Nov 21. PMID 21104112
- [Background] Virkki R, Juven T, Rikalainen H, Svedstrom E, Mertsola J, Ruuskanen O. Differentiation of bacterial and viral pneumonia in children. Thorax. 2002 May;57(5):438-41. doi: 10.1136/thorax.57.5.438. PMID 11978922
- [Background] Jain S, Williams DJ, Arnold SR, Ampofo K, Bramley AM, Reed C, Stockmann C, Anderson EJ, Grijalva CG, Self WH, Zhu Y, Patel A, Hymas W, Chappell JD, Kaufman RA, Kan JH, Dansie D, Lenny N, Hillyard DR, Haynes LM, Levine M, Lindstrom S, Winchell JM, Katz JM, Erdman D, Schneider E, Hicks LA, Wunderink RG, Edwards KM, Pavia AT, McCullers JA, Finelli L; CDC EPIC Study Team. Community-acquired pneumonia requiring hospitalization among U.S. children. N Engl J Med. 2015 Feb 26;372(9):835-45. doi: 10.1056/NEJMoa1405870. PMID 25714161
- [Background] Zar HJ, Barnett W, Stadler A, Gardner-Lubbe S, Myer L, Nicol MP. Aetiology of childhood pneumonia in a well vaccinated South African birth cohort: a nested case-control study of the Drakenstein Child Health Study. Lancet Respir Med. 2016 Jun;4(6):463-72. doi: 10.1016/S2213-2600(16)00096-5. Epub 2016 Apr 21. PMID 27117547
- [Background] Berkley JA, Munywoki P, Ngama M, Kazungu S, Abwao J, Bett A, Lassauniere R, Kresfelder T, Cane PA, Venter M, Scott JA, Nokes DJ. Viral etiology of severe pneumonia among Kenyan infants and children. JAMA. 2010 May 26;303(20):2051-7. doi: 10.1001/jama.2010.675. PMID 20501927
- [Background] Spichak TV, Yatsyshina SB, capital KA, Cyrillicatosova Lcapital KA, Cyrillic, capital KA, Cyrillicim SS, Korppi MO. Is the role of rhinoviruses as causative agents of pediatric community-acquired pneumonia over-estimated? Eur J Pediatr. 2016 Dec;175(12):1951-1958. doi: 10.1007/s00431-016-2791-x. Epub 2016 Oct 6. PMID 27714467
- [Background] van Gageldonk-Lafeber AB, Heijnen ML, Bartelds AI, Peters MF, van der Plas SM, Wilbrink B. A case-control study of acute respiratory tract infection in general practice patients in The Netherlands. Clin Infect Dis. 2005 Aug 15;41(4):490-7. doi: 10.1086/431982. Epub 2005 Jul 15. PMID 16028157
- [Background] Loeffelholz MJ, Trujillo R, Pyles RB, Miller AL, Alvarez-Fernandez P, Pong DL, Chonmaitree T. Duration of rhinovirus shedding in the upper respiratory tract in the first year of life. Pediatrics. 2014 Dec;134(6):1144-50. doi: 10.1542/peds.2014-2132. Epub 2014 Nov 17. PMID 25404719
- [Background] Chonmaitree T, Alvarez-Fernandez P, Jennings K, Trujillo R, Marom T, Loeffelholz MJ, Miller AL, McCormick DP, Patel JA, Pyles RB. Symptomatic and asymptomatic respiratory viral infections in the first year of life: association with acute otitis media development. Clin Infect Dis. 2015 Jan 1;60(1):1-9. doi: 10.1093/cid/ciu714. Epub 2014 Sep 9. PMID 25205769
- [Background] Spuesens EB, Fraaij PL, Visser EG, Hoogenboezem T, Hop WC, van Adrichem LN, Weber F, Moll HA, Broekman B, Berger MY, van Rijsoort-Vos T, van Belkum A, Schutten M, Pas SD, Osterhaus AD, Hartwig NG, Vink C, van Rossum AM. Carriage of Mycoplasma pneumoniae in the upper respiratory tract of symptomatic and asymptomatic children: an observational study. PLoS Med. 2013;10(5):e1001444. doi: 10.1371/journal.pmed.1001444. Epub 2013 May 14. PMID 23690754
- [Background] Chen SP, Huang YC, Chiu CH, Wong KS, Huang YL, Huang CG, Tsao KC, Lin TY. Clinical features of radiologically confirmed pneumonia due to adenovirus in children. J Clin Virol. 2013 Jan;56(1):7-12. doi: 10.1016/j.jcv.2012.08.021. Epub 2012 Sep 26. PMID 23021965
- [Background] Ortqvist AK, Lundholm C, Wettermark B, Ludvigsson JF, Ye W, Almqvist C. Validation of asthma and eczema in population-based Swedish drug and patient registers. Pharmacoepidemiol Drug Saf. 2013 Aug;22(8):850-60. doi: 10.1002/pds.3465. Epub 2013 Jun 11. PMID 23754713
- [Derived] Eklundh A, Rhedin S, Peltola V, Waris M, Naucler P, Gaudenzi G, Iacobelli A, Lindh M, Andersson M, Martensson A, Alfven T, Ryd-Rinder M. Evaluation of the Antigen mariPOC Respi Test Versus PCR in Relation to Immunological Viral Response in Children With Lower Respiratory Tract Infection. Int J Microbiol. 2025 Oct 15;2025:8832419. doi: 10.1155/ijm/8832419. eCollection 2025. PMID 41132494